CLINICAL TRIAL: NCT06178432
Title: A Single-arm, Open-label, Single-dose Study to Evaluate the Safety, Tolerability, and Efficacy of CRG003 Injection in the Treatment of Late Onset Pompe Disease
Brief Title: Evaluation of the Safety, Tolerability and Efficacy of Gene Therapy Drug for Late Onset Pompe Disease (LOPD)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, MD, PhD, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2023-783
Record Dates: First submitted 2023-11-30; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Pompe Disease (Late-onset)
Keywords: LOPD
MeSH Terms: conditions — Glycogen Storage Disease Type II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm of CRG003 injection (Experimental): The dose of CRG003 injection will be calculated according to the participant's weight with single intravenous infusion.
  Interventions: Genetic: CRG003 injection

INTERVENTIONS:
Genetic: CRG003 injection — The dose of CRG003 will be calculated according to the participant's weight with single intravenous infusion.
  Other Names: BBM-G102 injection

SUMMARY:
This is a single-center, single-arm, open-label, single-dose treatment clinical study to evaluate the safety, tolerability and efficacy of CRG003 injection in participants with late onset Pompe disease (LOPD), with a long-term follow-up period of 5 years.

CRG003 (BBM-G102) injection is an adeno-associated virus (AAV) gene therapy product for treating Pompe disease to stably express active GAA enzyme in the liver on a long-term basis after the injection.

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily sign informed consent form;
2. Clinically diagnosed with LOPD;
3. Males or females aged ≥ 18 years;
4. Undergone enzyme replacement treatment (ERT) with recombinant human acid alpha-glucosidase (rhGAA) previously, and has been discontinued for at least four weeks before screening;
5. Acceptable Pulmonary test results;
6. A 6MWT ≥ 100 meters, and ambulation for 40 meters without stopping and without an assistive device;
7. Acceptable laboratory values;
8. Acceptable GAA anti-drug antibody titer;
9. Acceptable capsid antibody titers;
10. Use of reliable contraception methods during the study;
11. Participants with good compliance.

Exclusion Criteria:

1. Severe cardiomyopathy was defined as left ventricular ejection fraction (LVEF) < 45% or New York Heart Association (NYHA) functional class 3 or above;
2. Require invasive mechanical ventilation, or rely on noninvasive ventilation during the day;
3. Intolerance to ERT, prior experience of serious infusion-associated reactions (IARs), prior experience of serious allergic reactions or investigator-assessed intolerance to ERT;
4. Have received any systemic immunosuppressants (except inhalation or topical use) other than glucocorticoids or investigator-recommended immunosuppressants 30 days prior to screening, and known intolerance to immunosuppressants such as glucocorticoids;
5. Positive for hepatitis B surface antigen (HBsAg) or hepatitis B virus DNA (HBV-DNA), positive for hepatitis C virus RNA (HCV-RNA). Participants with a history of hepatitis B or C can be regarded as negative if both two samples collected at an interval of at least three months are tested negative for the above parameters; positive for human immunodeficiency virus (HIV) or positive serologic test for syphilis;
6. Currently on antiviral therapy for hepatitis B or C;
7. Have clinical organic diseases (except symptoms or diseases associated with Pompe disease), including active tuberculosis, cardiovascular and cerebrovascular diseases, hepatobiliary system, respiratory system, nervous system, urinary system, or endocrine system disorders (such as diabetes, etc.), or other serious complications, or other conditions that make the patients not eligible for the study according to the investigator;
8. Have underlying liver diseases, e.g., prior diagnosis of portal hypertension, splenomegaly, hepatic encephalopathy, severe fatty liver, cirrhosis or liver fibrosis ≥stage 3; or ultrasound-identified liver neoplasms or laboratory tests suggesting elevated alpha-fetoprotein, etc., which are considered by the investigator as clinically significant;
9. Have received gene therapy prior to screening or used other investigational drugs or drugs that affect this study as evaluated by the investigator within four weeks prior to screening or within 5 half lives of the investigational drug (whichever is longer);
10. Have received or will receive any herbal preparations (herbal supplements or traditional Chinese medicines derived from plants, minerals, or animals, other than topical medications) that may affect liver function or Chinese herbal medicines that may affect the study as judged by the investigator four weeks prior to study medication or during the study follow-up period;
11. Alcohol dependence or drug addiction, and inability to stop alcohol intake as ordered by the doctor during the study;
12. Have received any live vaccine two months predose or history of vaccination within 30 days prior to screening or planning to receive vaccination during the screening and the main study period;
13. Pregnant or lactating female participants;
14. Other conditions that make the participants not eligible for the study according to the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limited toxicities | 12 weeks
  Incidence of dose limited toxicities (DLTs) as determined by the safety review committee (SRC) within 12 weeks following CRG003 infusion;
Incidence of adverse events and serious adverse events | 26 weeks and 52 weeks
  Incidence of adverse events (AEs) and serious adverse events (SAEs) within 26 weeks and 52 weeks following CRG003 infusion
The change of hepatic enzyme concentration | 26 weeks and 52 weeks
  Alkaline phosphatase (ALP)
Changes from baseline in liver function | 26 weeks and 52 weeks
  Changes from baseline in liver function [Alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT) and total bilirubin (TBIL)] within 26 weeks and 52 weeks following CRG003 infusion

CONTACTS AND LOCATIONS:
Overall Officials: Chongbo Zhao, MD,PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No